CLINICAL TRIAL: NCT00780520
Title: The Effect of Glutamine Infusion on the Inflammatory Response and HSP-70 in BMNCs During Human Experimental
Brief Title: The Effect of Glutamine on Systemic Inflammation During Human Experimental Endotoxemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: H-KF-01-144/98
Record Dates: First submitted 2008-10-24; First posted 2008-10-27 (Estimated); Last update posted 2008-10-27 (Estimated); Status verified 2008-10

CONDITIONS: Sepsis; Systemic Inflammation
Keywords: glutamine inflammation HSP70 sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Dietary Supplement: alanine-glutamine infusion
- 2 (Placebo Comparator)
  Interventions: Dietary Supplement: alanine-glutamine infusion

INTERVENTIONS:
Dietary Supplement: alanine-glutamine infusion

SUMMARY:
Glutamine levels decrease during severe sepsis; this may be associated with increased mortality. The investigators tested the effects of glutamine supplementation on systemic inflammation in a human sepsis model.

The investigators found that glutamine levels drops significantly during experimentally induced systemic inflammation. However, glutamine did not affect the degree of inflammation.

DETAILED DESCRIPTION:
Glutamine levels have been shown to decrease substantially with severe sepsis and this has been connected with increased mortality. Therefore, in the present study, we infused either saline or Alanine-glutamine during an endotoxin challenge and measured parameters related to an immune response, i.e. plasma cytokines and Heat Shock Protein (HSP)-70.

Materials and Methods This was a double blind, randomised, placebo-controlled crossover trial in eight healthy young men. The study was performed in random order on two separate days, with a four-week washout period between days. Subjects received an infusion of Alanine-glutamine ( Dipeptiven) at a rate of 0.025 g / (kg BW * h) for 10 hrs or saline. After two hours of infusion subjects received an intravenous bolus of E. coli endotoxin (0.3 ng/kg). Blood samples were collected hourly for the following eight hours. HSP-70 protein content in isolated Blood Mononuclear Cells (BMNCs) was measured by western blotting.

Results and Discussion Plasma glutamine was significantly increased during infusion with alanine-glutamine infusion. En-dotoxin caused a reduction in plasma-glutamine during saline infusion as well as during Alanine-glutamine infusion. A significant effect of endotoxin was found on leukocyte subpopulations, tumor necrosis factor-a, interleukin-6, the expression of HSP-70 in BMNCs, temperature, and heart rate. However, no differences were detected between treatments with regard to the effect of endotoxin on any of these parameters.

Conclusion Endotoxemia reduces plasma glutamine independently of parenteral infusion of alanine-glutamine. Glutamine does not alter the response of leukocytes, leukocyte subpopulations, IL-6, or TNF-α, or the expression of HSP-70 in BMNCs to endotoxemia.

ELIGIBILITY:
Inclusion Criteria:

* Healthy young males

Exclusion Criteria:

* Any kind of acute or chronic diseases

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2007-06; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Plasma-levels of cytokines

SECONDARY OUTCOMES:
Heat shock protein -70 production from BMNCs

CONTACTS AND LOCATIONS:
Locations (1):
- Centre of Inflammation and Metabolism, Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Derived] Andreasen AS, Pedersen-Skovsgaard T, Mortensen OH, van Hall G, Moseley PL, Pedersen BK. The effect of glutamine infusion on the inflammatory response and HSP70 during human experimental endotoxaemia. Crit Care. 2009;13(1):R7. doi: 10.1186/cc7696. Epub 2009 Jan 27. PMID 19173710